CLINICAL TRIAL: NCT07065942
Title: Effects of Lactulose on Gut Microbiota and Metabolism in Diabetic Constipated Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Beijing Hospital (Other Government); Beijing Huaxin Hospital (Unknown); Beijing Luhe Hospital (Other); Beijing Huairou Hospital (Other)
Responsible Party: Principal Investigator, Jing-Nan Li, Chief physician, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I-23PJ993
Record Dates: First submitted 2025-07-04; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-06

CONDITIONS: Diabetes Mellitus; Constipation - Functional
Keywords: Diabetes; Constipation; Lactulose; Gut Microbiota; Metabolism
MeSH Terms: conditions — Diabetes Mellitus; Constipation | interventions — Lactulose

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lactulose Oral Solution (Active Comparator)
  Interventions: Drug: Lactulose oral solution
- Lactulose Oral Solution+Live Combined B. Subtilis and E. Faecium Enteric-coated Capsules (Experimental)
  Interventions: Drug: Lactulose oral solution; Drug: Live Combined B. Subtilis and E. Faecium Enteric-coated Capsules

INTERVENTIONS:
Drug: Lactulose oral solution — Oral, 30 mL once daily administered during breakfast.
Drug: Live Combined B. Subtilis and E. Faecium Enteric-coated Capsules — Oral, 2 tablets (500 mg per tablet) three times daily (TID).
  Arms: Lactulose Oral Solution+Live Combined B. Subtilis and E. Faecium Enteric-coated Capsules

SUMMARY:
Constipation is the most common gastrointestinal manifestation in diabetic patients. Emerging evidence suggests that gut microbiota dysbiosis may contribute to the pathogenesis of diabetes, highlighting the need to investigate its role in diabetic constipation, though current research remains limited.

Current management of diabetic constipation primarily relies on bulk-forming and osmotic laxatives. Additionally, microbiome-modulating agents (e.g., probiotics, prebiotics, and synbiotics) may serve as adjunctive therapies by regulating gut microbiota and enhancing intestinal motility. Lactulose, a well-tolerated osmotic laxative with prebiotic effects, is widely recommended in clinical guidelines. It promotes short-chain fatty acid production, increases fecal volume, and accelerates colonic transit, thereby alleviating constipation. However, its specific impact on gut microbiota composition and metabolic pathways in diabetic constipation remains unclear.

This study aims to explore changes in fecal microbiota and metabolomic profiles in diabetic patients with chronic constipation following treatment with lactulose alone or in combination with Bacillus subtilis-Enterococcus faecium probiotics, providing mechanistic insights into prebiotic therapy for this condition.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-70 years
* Type 2 Diabetes Diagnosis (per 2017 ADA criteria), meeting ≥1 of:

  1. Fasting plasma glucose (FPG) ≥7.0 mmol/L
  2. hour plasma glucose ≥11.1 mmol/L during 75g anhydrous oral glucose tolerance test (OGTT)
  3. Random plasma glucose ≥11.1 mmol/L with hyperglycemia symptoms or hyperglycemic crisis
* Functional Constipation (Rome IV criteria), requiring:

  1. ≥2 of the following

     1. occurring in ≥25% of defecations
     2. Straining
     3. Lumpy/hard stools (Bristol Stool Scale 1-2)
     4. Sensation of incomplete evacuation
     5. Anorectal obstruction/blockage
     6. Manual maneuvers required
     7. <3 spontaneous bowel movements/week
  2. No loose stools without laxatives
  3. Exclusion of IBS diagnosis. Symptom duration >6 months, with active symptoms meeting criteria for last 3 months.
* Stable Glycemic Control: No anticipated antidiabetic medication adjustments during study
* Dietary Stability: Maintain consistent diet; avoid yogurt, fermented foods, prebiotic-containing processed foods, or other items that may confound results

Exclusion Criteria:

* Secondary Constipation due to organic diseases or medication effects.
* Constipation-predominant Irritable Bowel Syndrome (IBS-C).
* Concurrent gastrointestinal disorders (e.g., inflammatory bowel disease, colorectal cancer).
* Type 1 Diabetes Mellitus.
* Severe chronic comorbidities, including:

  1. Cardiopulmonary insufficiency
  2. Cerebrovascular diseases
  3. Psychiatric disorders
* Recent use (within 1 month) of confounding medications:

  1. Probiotics/prebiotics
  2. Antibiotics
  3. Laxatives (e.g., osmotic/stimulant agents)
  4. Prokinetics

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Changes in Constipation Symptom Scores Pre- and Post-Treatment | From enrollment (0 week) to 2 weeks, and 4 Weeks at the end of treatment
  Assessment of treatment efficacy on constipation symptoms: Changes in symptom scores from baseline to post-treatment within each treatment arm and comparative analysis between the lactulose monotherapy group and lactulose+Medilac-S combination therapy group
Changes in Fecal Microbiota Composition (16S rRNA and Metagenomics) | From enrollment (0 week) to 2 weeks, and 4 Weeks at the end of treatment
  Comparison of Fecal Microbiota Composition Changes (16S rRNA and Metagenomics): Pre- vs. Post-Treatment Alterations and Intergroup Differences Between Lactulose Monotherapy and Lactulose+Medilac-S Combination Therapy
Temporal Changes in Fecal Untargeted Metabolomics Profiles | From enrollment (0 week) to 2 weeks, and 4 Weeks at the end of treatment
  Temporal Changes in Fecal Untargeted Metabolomics Profiles: Pre- vs. post-treatment alterations and comparative analysis between lactulose monotherapy and lactulose+Medilac-S combination groups.

SECONDARY OUTCOMES:
Changes in Fasting Blood Glucose and Glycated Albumin Levels | From enrollment (0 week) to 2 weeks, and 4 Weeks at the end of treatment
  Changes in Fasting Blood Glucose and Glycated Albumin Levels: Pre- vs. post-treatment variations and comparative analysis between lactulose monotherapy and lactulose+Medilac-S combination groups
Changes in Blood Lipid Profiles (Total Cholesterol, Triglycerides, HDL-C, and LDL-C) | From enrollment (0 week) to 2 weeks, and 4 Weeks at the end of treatment
  Changes in Blood Lipid Profiles (Total Cholesterol, Triglycerides, HDL-C, and LDL-C): Pre- vs. post-treatment alterations and comparative analysis between lactulose monotherapy and lactulose+Medilac-S combination therapy groups

CONTACTS AND LOCATIONS:
Overall Officials: Jingnan Li, MD, Ph.D, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No